CLINICAL TRIAL: NCT03142269
Title: The Influences of 360° Anterior Capsule Polishing on Refraction, Anterior Capsular Opening Size and IOL Stability Among Super High Myopia Patients
Brief Title: The Influences Of Anterior Capsule Polishing On Anterior Capsular Changes and Intraocular Lenses Stability of Super High Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: yin ying zhao (Other)
Responsible Party: Sponsor-Investigator, yin ying zhao, doctor, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: kyk201601
Record Dates: First submitted 2017-02-25; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Myopia, High, With Cataract and Anterior Capsule Polished
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polished group (Active Comparator): 360°anterior capsule polishing was performed with double-ended capsule polisher randomly in one eye
  Interventions: Procedure: 360°anterior capsule polishing
- unpolished group (Placebo Comparator): the opposite unpolished was used as the control
  Interventions: Procedure: 360°anterior capsule polishing

INTERVENTIONS:
Procedure: 360°anterior capsule polishing — 360°anterior capsule polishing was performed with double-ended capsule polisher

SUMMARY:
A prospective study included 20 patients with super high myopia who underwent bilateral uneventful cataract. 360°anterior capsule polishing was performed with double-ended capsule polisher randomly in one eye, and the opposite unpolished was used as the control. The refractive state and size of anterior opening were measured at postoperative 1 day as the baseline. Then they followed up at 1 month, 3 months and 6 months after surgery to record refractive state, higher-order aberrations, size of anterior opening, tilt and decentration of IOL (intraocular lenses)and PAD(postoperative aqueous depth). The paired t test was used to compare the differences between the two groups, and the same test the postoperative follow-up comparing with the baseline.

ELIGIBILITY:
Inclusion Criteria:cataract patients with super high myopia (axial length >27mm) and difference of binocular was less than 1mm Exclusion Criteria:larger corneal astigmatism need toric intraocular lens; patients with any systemic or ocular diseases that may influence the anterior capsule opening morphologic, such as keratonosus, glaucoma, uveitis, Pseudoexfoliation syndrome, retinitis pigmentosa and diabetes and Myotonic Dystrophy, etc.; patients with ophthalmic surgery and trauma history.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
refraction | Change from postoperative 1 day to 1 months
  refractive state
anterior opening size | Change from postoperative 1 day to 1 months
  area,diameter
Stability of IOL | Change from postoperative 1 months to 3 months
  Tilt and Decentration

SECONDARY OUTCOMES:
refraction | Change from postoperative 1 month to 3 months
  refractive state
refraction | Change from postoperative 3 month to 6 months
  refractive state
anterior opening size | Change from postoperative 1 month to 3 months
  area,diameter
anterior opening size | Change from postoperative 3 month to 6 months
  area,diameter
Stability of IOL | Change from postoperative 3 month to 6 months
  Tilt and Decentration